CLINICAL TRIAL: NCT05233605
Title: Impact of Post-ARDS Covid Sedation on Persistent Neuroinflammation (PET-DEXDOCOVID)
Brief Title: Impact of Post-ARDS Covid-19 Sedation on Persistent Neuroinflammation
Acronym: PET-DEXDOCOVID
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200491; 2020-004802-70 (EudraCT Number)
Record Dates: First submitted 2021-10-15; First posted 2022-02-10 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Severe COVID-19
Keywords: SARS-Cov 2 (Severe Acute Respiratory Syndrome-Coronavirus 2); Covid-19; Dexmedetomidine; Neuroinflammation; [18F]-DPA-714; PET-MRI
MeSH Terms: conditions — COVID-19; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples (serum, blood mononuclear cells, total proteins for cytof, transcriptome and epigenome) will constitute biological collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposed to Dexmedetomidine during ICU stay: Dexmedetomidine has been administered in accordance with its MA (at least 24 hours continuously with a starting dose of 0.7 µg/kg/h and then adjusted to sedation scores between 0.4 and 1.1 µg/kg/h), as part of care, prior to inclusion in the protocol
- Not Exposed to Dexmedetomidine during ICU stay: Standard of care

SUMMARY:
ICU Patients admitted after ARDS due to COVID infection should be weaned from invasive mechanical ventilation as quickly as possible.

60% of ARDS patient after COVID infection admitted in ICU developp a delirium during mechanical ventilation weaning, serious event that can lead to death or acute and late complications since 30% of patients who had a delirium in ICU develop cognitive sequelae. Based on epidemiological arguments and mouse models, severe neuroinflammation is considered to be one of the physiopathological mechanisms causing delirium during ventilatory weaning.

In addition to its sedative properties, dexmedetomidine exhibits neuroprotective effects. In experimental models, dexmedetomidine reduces brain inflammation acting directly on the microglial phenotype. The role of this chronic neuroinflammatory condition on cognitive abilities and reserve begins to emerge in the literature no matter the initial stress is (surgery, head trauma, or Alzheimer's type dementia) and is therefore able to influence quality of life. The evaluation of this neuroinflammation by non-invasive tools appears essential in the management and follow-up of post-COVID cerebrolesed patients, as well as the potentially neuroprotective evaluation of dexmedetomidine.

DETAILED DESCRIPTION:
COVID-19 is responsible of a pandemic since December 31 2019, which began in China and spread rapidly. Confirmed Covid positive patients worlwide is estimated at 179 M in June 2021. The infection started in France at the beginning of 2020 and causes severe pneumonia with 130,519 confirmed cases, including 2,712 (2.1%) hospitalizations in intensive care units. COVID-19 emerges as a poorly understood systemic disease that affects several organs, especially the lungs. The first reason for worsening and hospitalization in intensive care is acute respiratory distress syndrome (ARDS) that requires heavy and long care management with orotracheal intubation and mechanical ventilation, as well as prolonged sedation and curarization. Patients who survived this critical phase should then be weaned from this invasive monitoring as quickly as possible to limit risk of morbidity and mortality. It therefore appears essential to do everything possible to reduce the duration of mechanical ventilation and the period of ventilatory weaning, a real daily challenge in intensive care, for both medical and socio-economic sides.

Beside COVID-19 infection, the ventilatory weaning phase is a long and difficult period that can last more than 40 to 60% of the time spent under mechanical ventilation and can be more complicated as the duration of sedation is prolonged. This phase is correlated with the duration of mechanical ventilation, as well as with respiratory, cardiac and neuromuscular diseases. Considering all the risk factors for prolonged ventilatory weaning, one of these is the intensive care delirium.

Delirium in intensive care is a serious event, possibly leading to mortality or acute and late complications (self-extubation, catheter removal, ...) since 30% of delirium patients develop cognitive sequelae. The incidence of this post-ARDS delirium is approximately 20% according to the studies and is found predominantly in patients with severe sepsis. The academic tool to access delirium in intensive care is the CAM-ICU (Confusion Assessment Mehod - ICU) scale; the RASS score (Richmond Agitation-Sedation Scale) is also usable to access patients with a hyperactive form (RASS score greater than 2).

Several drug strategies based on the use of sedating agents such as dexmedetomidine or certain neuroleptics such as loxapine or haloperidol have been developed to reduce this incidence. Dexmedetomidine is a selective adrenergic receptor agonist and has hypnotic and analgesic properties.

At the same time, dexmedetomidine exhibits neuroprotective effects. In experimental models such as intraperitoneal injection of lipopolysaccharide or LPS, marrow lesions or ischemia-reperfusion models, dexmedetomidine reduces cerebral inflammation with a direct action on the microglial phenotype. The impacted signaling pathway is still unclear, however several studies show an action of dexmedetomidine on the AMPK pathway. The use of dexmedetomidine to prevent and treat delirium is not uniform within intensive care units in France and is not administered systematically.

Unexpectedly, two thirds of patients hospitalized in intensive care for ARDS after COVID-19 infection develop a severe delirium. This unique incidence is double the incidences found in other populations in ICU (sepsis, meningitis,...).

Neuroinflammation reaction induced by an intra or extra-cranial phenomenon is a very studied process.

The latter is totally correlated with the strength of the stimulus and can be the cause of a disturbance or a complete runaway of the immune system described in the literature as an inflammatory storm. This neuroinflammation induced during the IC hospitalization is now known to persist, until several years after outbreak.

The role of this chronic neuroinflammatory persistent response on cognitive capacities and reserve begins to emerge in the literature regardless of the initial stress (surgery, head trauma, or Alzheimer-type dementia) and is therefore capable of influencing the quality of life of patients. The evaluation of this neuroinflammation using non-invasive tools appears to be essential in the management of cerebrolesed patients.

Among existing tools, positron emission tomography (PET) imaging using radiotracers specific for monocytic/microglial activation is now recognized as a relevant tool because of its sensitive and specific characteristics to assess brain inflammation. Several radiotracers have been tested, in particular [11C] -PK11195, but it is [18F] -DPA-714 or DPA that is retained in the literature because it has many pharmacokinetic advantages. He has indeed shown his interest in a few animal and human models in various pathologies. It should be noted that the DPA receptor exhibits a polymorphism that may explain certain differences in binding observed in humans. This tool, by means of a quantitative and possibly regional measurement of the signal measurement, is particularly innovative and seems to correlate with cognitive disorders, particularly in the context of Alzheimer's disease. Currently, the technology combining MRI and PET imaging with DPA appears to be the most successful for evaluating neuroinflammation, allowing regional measurement with better resolution. Recent studies have also been able to show that the increase in DPA by PET-MRI was associated with a pejorative cognitive evolution.

The role of peripheral inflammation on the neuro-inflammatory profile is now well described with both mediation via cytokines / chemokines produced by systemic immunity but also by infiltration and cellular exchanges of the monocyte / macrophage cells, which interact directly with the microglia. Although the full range of mechanisms is still poorly understood, it seems that there is a very close communication between the peripheral immune system and the central nervous system, causing an initial inflammatory runaway. Thus, it seems opportune in our cohort for which neuroinflammation is suspected, to combine the quantification of the main circulating mediators (cytokine and chemokine assays) and cellular (PBMC cell sorting [Peripheral blood mononuclear cells], with transcriptomic and epigenomic analysis as well as proteomics with time-of-flight cytometry or Cytof) easily accessible in the blood of patients in order to best describe in a minimally invasive manner this inflammatory reaction and to be able propose a follow-up and a potential therapeutic strategy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥ 18 years at the time of inclusion) under 75 years old
* COVID-19 infection documented by PCR test performed on a nasopharyngeal swab or from a bronchoalveolar sample
* High affinity homozygous TPSO genotyping for [18F] -DPA-714 or heterozygous intermediate affinity for [18F] -DPA-714
* Patient who was hospitalized in intensive care for ARDS after COVID infection which required mechanical ventilation and deep sedation for at least 24 hours
* Patient alive at 24 months (+ 24 months) after discharge from intensive care
* Signature of informed consent
* Patient affiliated to a National French social security system, excluding (French) State Medical Aid (SMA)

For the group of patients exposed to dexmedetomidine:

* Administration of dexmedetomidine for at least 24 hours during intensive care hospitalization

For the group of patients not exposed to dexmedetomidine:

* No administration of dexmedetomidine during intensive care hospitalization

Exclusion Criteria:

* Protected adult (under legal protection, guardianship or curatorship)
* Pregnancy or breast-feeding
* Contraindication to PET or MRI examination
* Severe renal impairment (creatinine clearance <30 mL / min)
* Contraindication to the administration of the radiopharmaceutical agent [18F]-DPA-714
* Serious neurological history at admission to intensive care:

  * Stroke
  * Severe head trauma
  * Dementia with loss of autonomy

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted in ICU for COVID-19 ARDS and alive 2 years after infection
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
Mean of SUVr of [18F]-DPA-714 in frontal lobes compared to cerebellar lobes | 24 months (+ 24 months) after ICU discharge
  Persistent neuroinflammation is measured by [18F]-DPA-714 signal intensity obtained on PET-MRI imaging on the 2 frontal lobes (freesurfer segmentation, with signal intensity being the ratio of the measurement in the frontal lobes to that in the cerebellar lobes. The standard fixation will be expressed as an indexed value compared to the control value.
  The intensity of the [18F]-DPA-714 signal is the SUV (standard uptake value) or quantity of radioactivity fixed in the tissue which will be measured in each region of interest (frontal lobes and cerebellar lobes = reference) and related to the quantity of radioactivity injected for the examination.
  This signal will be corrected by taking into account the weight, the amount of radioactivity injected for the examination and the SNPrs6971 genotype (low, medium or high affinity of the radiotracer for its ligand).
  The ratio of SUV in the frontal lobes to the SUV of the cerebellar lobes

SECONDARY OUTCOMES:
Neuro-cognitive lesions acquired using clinical assessment score means | 24 months (+24 months) after ICU discharge
  Neuro-cognitive lesions acquired using clinical assessment score GOSE
Neuro-cognitive lesions acquired using clinical assessment score means | 24 months (+24 months) after ICU discharge
  Neuro-cognitive lesions acquired using clinical assessment score Rankin
Neuro-cognitive lesions acquired using clinical assessment score means | 24 months (+24 months) after ICU discharge
  Neuro-cognitive lesions acquired using clinical assessment score: presence of memory impairment assessed by MOCA
Neuro-cognitive lesions acquired using clinical assessment score means | 24 months (+24 months) after ICU discharge
  Neuro-cognitive lesions acquired using clinical assessment score: presence of memory impairment assessed by GOAT score
Neuro-cognitive lesions acquired using clinical assessment score means | 24 months (+24 months) after ICU discharge
  Neuro-cognitive lesions acquired using clinical assessment score: presence of depressive state by HADS
Neuro-cognitive lesions acquired using clinical assessment score means | 24 months (+24 months) after ICU discharge
  Neuro-cognitive lesions acquired using clinical assessment score: dependencies by the Barthel score
Neuro-cognitive lesions acquired using clinical assessment score means | 24 months (+24 months) after ICU discharge
  Neuro-cognitive lesions acquired using clinical assessment score: presence of a PTSD
Neuro-cognitive lesions acquired using clinical assessment score means | 24 months (+24 months) after ICU discharge
  Neuro-cognitive lesions acquired using clinical assessment score: the quality of life scale SF36
Neuro-cognitive lesions acquired using clinical assessment score means | 24 months (+24 months) after ICU discharge
  Neuro-cognitive lesions acquired using clinical assessment score Qolibri
Neuro-cognitive lesions acquired using clinical assessment score means | 24 months (+24 months) after ICU discharge
  Neuro-cognitive lesions acquired using clinical assessment score GDS
Neuro-cognitive lesions acquired using clinical assessment score means | 24 months (+24 months) after ICU discharge
  Neuro-cognitive lesions acquired using clinical assessment score: detection of anorexia by the DSM-IV-TR scale and DSM-V.
Neuro-cognitive lesions acquired using clinical assessment score means | 24 months (+24 months) after ICU discharge
  Neuro-cognitive lesions acquired using clinical assessment score: detection of anorexia by the DSM-V
Mean of neuro-cognitive lesions acquired using diffusion tensor brain MRI | 24 months (+24 months) after ICU discharge
  Neuro-cognitive lesions acquired using diffusion tensor brain MRI will be documented by: overall brain volume, brain volume in certain regions (corpus callosum, thalami, cerebrospinal fluid, cerebellum), and an assessment of white matter lesions (measurement of the anisotropy fraction (FA), mean diffusivity (MD), L1 and Lt) and this also at the level of the overall brain and in certain regions precisely.
Study the distribution of SUVr in different freesurfer regions on the PET-MRI examination | 24 months (+24 months) of discharge from intensive care
  DPA signal will be quantified in each ROIs and will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent DEGOS, Pr, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Anesthesy department - Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.